CLINICAL TRIAL: NCT00740454
Title: Diagnostic Exclusion Value of a Negative Single Distal and Proximal Lower Limb Veins Compression Ultrasonography in Pregnant and Post-partum Women With a Clinically Suspected Deep Vein Thrombosis
Brief Title: Single Complete Compression Ultrasonography to Rule Out Deep Vein Thrombosis During Pregnancy and Postpartum
Acronym: EDVIGE
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: EDVIGE
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Deep Vein Thrombosis
Keywords: pregnancy; postpartum; deep vein thrombosis; venous thromboembolism; diagnosis; compression ultrasonography
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Pregnant or post-partum women with a clinically suspected DVT and a negative distal and proximal leg veins compression ultrasonography
  Interventions: Other: Lower limb veins compression ultrasonography

INTERVENTIONS:
Other: Lower limb veins compression ultrasonography — Distal and proximal lower limb veins compression ultrasonography

SUMMARY:
The objective of the EDVIGE study is to determine whether a negative single distal and proximal leg veins compression ultrasonography safely rules out the diagnosis of deep vein thrombosis in pregnant and post-partum women with clinical suspicion of DVT.

DETAILED DESCRIPTION:
A single distal and proximal leg veins compression ultrasonography has been shown to safely rule out the diagnosis of DVT when negative. The safety of this strategy has never been verified in pregnant or postpartum women. It could however be limited in that clinical setting, because of modified hemodynamics, hampered observation conditions, lack of respiratory modulation, higher proportion of isolated iliac deep vein thromboses. The objective of the EDVIGE study is to assess the safety of this diagnostic strategy during pregnancy and post-partum.

ELIGIBILITY:
Inclusion Criteria:

* Women with an ongoing pregnancy or within three-months post-partum and a clinically suspected deep vein thrombosis

Exclusion Criteria:

* suspicion of pulmonary embolism
* age less than 18 years
* impossible follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant or post-partum women referred to primary care vascular medicine physicians or diagnostic imaging units of referral hospitals in Brittany (France) and Geneva (Switzerland)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2006-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Objectively confirmed thromboembolic events | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregoire LE GAL, MD, PhD, Principal Investigator — Brest University Hospital, Brest, France
Locations (2):
- EA3878, Brest University Hospital, Brest, France
- Division of Angiology and Hemostasis, Geneva University Hospital, Geneva, Switzerland

REFERENCES:
- [Background] Le Gal G, Prins AM, Righini M, Bohec C, Lacut K, Germain P, Vergos JC, Kaczmarek R, Guias B, Collet M, Bressollette L, Oger E, Mottier D. Diagnostic value of a negative single complete compression ultrasound of the lower limbs to exclude the diagnosis of deep venous thrombosis in pregnant or postpartum women: a retrospective hospital-based study. Thromb Res. 2006;118(6):691-7. doi: 10.1016/j.thromres.2005.12.004. Epub 2006 Jan 18. PMID 16414102
- [Derived] Righini M, Robert-Ebadi H, Cremonesi A, Elias A, Sanchez O, Le Moigne E, Schmidt J, Le Gall C, Cornuz J, Aujesky D, Roy PM, Chauleur C, Rouyer F, Poletti PA, Moreau C, Le Gal G; CT-PE-Pregnancy group. Risk of neonatal hypothyroidism in newborns from mothers exposed to CTPA during pregnancy: Ancillary data from a prospective outcome study. J Thromb Haemost. 2022 Nov;20(11):2550-2555. doi: 10.1111/jth.15843. Epub 2022 Aug 28. PMID 35950611
- [Derived] Righini M, Robert-Ebadi H, Elias A, Sanchez O, Le Moigne E, Schmidt J, Le Gall C, Cornuz J, Aujesky D, Roy PM, Chauleur C, Rutschmann OT, Poletti PA, Le Gal G; CT-PE-Pregnancy Group. Diagnosis of Pulmonary Embolism During Pregnancy: A Multicenter Prospective Management Outcome Study. Ann Intern Med. 2018 Dec 4;169(11):766-773. doi: 10.7326/M18-1670. Epub 2018 Oct 23. PMID 30357273
- [Derived] Righini M, Jobic C, Boehlen F, Broussaud J, Becker F, Jaffrelot M, Blondon M, Guias B, Le Gal G; EDVIGE study group. Predicting deep venous thrombosis in pregnancy: external validation of the LEFT clinical prediction rule. Haematologica. 2013 Apr;98(4):545-8. doi: 10.3324/haematol.2012.072009. Epub 2012 Oct 12. PMID 23065510
- [Derived] Le Gal G, Kercret G, Ben Yahmed K, Bressollette L, Robert-Ebadi H, Riberdy L, Louis P, Delluc A, Labalette ML, Baba-Ahmed M, Bounameaux H, Mottier D, Righini M; EDVIGE Study Group. Diagnostic value of single complete compression ultrasonography in pregnant and postpartum women with suspected deep vein thrombosis: prospective study. BMJ. 2012 Apr 24;344:e2635. doi: 10.1136/bmj.e2635. PMID 22531869